CLINICAL TRIAL: NCT02484547
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Aducanumab (BIIB037) in Subjects With Early Alzheimer's Disease
Brief Title: 221AD302 Phase 3 Study of Aducanumab (BIIB037) in Early Alzheimer's Disease
Acronym: EMERGE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued based on futility analysis done and not based on safety concerns. Follow-up visits and closing out study activities are completed
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221AD302; 2015-000967-15 (EudraCT Number)
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer's Disease
Keywords: Aducanumab; BIIB037
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Experimental): Monthly intravenous (IV) infusions
  Interventions: Drug: Aducanumab (BIIB037); Drug: Placebo
- High Dose (Experimental): Monthly intravenous (IV) infusions
  Interventions: Drug: Aducanumab (BIIB037); Drug: Placebo

INTERVENTIONS:
Drug: Aducanumab (BIIB037) — Low dose
  Arms: Low Dose
Drug: Aducanumab (BIIB037) — High dose
  Arms: High Dose
Drug: Placebo — Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of monthly doses of aducanumab in slowing cognitive and functional impairment as measured by changes in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) score as compared with placebo in participants with early AD. Secondary objectives are to assess the effect of monthly doses of aducanumab as compared with placebo on clinical progression as measured by Mini-Mental State Examination (MMSE), AD Assessment Scale-Cognitive Subscale (13 items) [ADAS-Cog 13], and AD Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment version) [ADCS-ADL-MCI].

ELIGIBILITY:
Key Inclusion Criteria:

* Must meet all of the following clinical criteria for MCI due to AD or mild AD and must have:
* A Clinical Dementia Rating (CDR)-Global Score of 0.5.
* Objective evidence of cognitive impairment at screening
* An MMSE score between 24 and 30 (inclusive)
* Must have a positive amyloid Positron Emission Tomography (PET) scan
* Must consent to apolipoprotein E (ApoE) genotyping
* If using drugs to treat symptoms related to AD, doses must be stable for at least 8 weeks prior to screening visit 1
* Must have a reliable informant or caregiver

Key Exclusion Criteria:

* Any medical or neurological condition (other than Alzheimer's Disease) that might be a contributing cause of the subject's cognitive impairment
* Have had a stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year
* Clinically significant unstable psychiatric illness in past 6 months
* History of unstable angina, myocardial infarction, advanced chronic heart failure, or clinically significant conduction abnormalities within 1 year prior to Screening
* Indication of impaired renal or liver function
* Have human immunodeficiency virus (HIV) infection
* Have a significant systematic illness or infection in past 30 days
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* Any contraindications to brain magnetic resonance imaging (MRI) or PET scans
* Alcohol or substance abuse in past 1 year
* Taking blood thinners (except for aspirin at a prophylactic dose or less)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1643 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (176):
- United States (58):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Xenoscience Inc., Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Institute for Memory Impairments, Irvine, California
  - Renewal Behavioral Health, Long Beach, California
  - USC Keck School of Medicine, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Excell Research, Inc., Oceanside, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Anderson Clinical Research, Redlands, California
  - Pacific Research Network, San Diego, California
  - University of California San Diego Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Stanford University Medical Center, Stanford, California
  - University Of Colorado Denver, Aurora, Colorado
  - IMMUNOe International Research Centers, Thornton, Colorado
  - Associated Neurologists of Southern Connecticut, PC, Fairfield, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Quantum Laboratories Inc., Deerfield Beach, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Emory University Cognitive Neurology Clinic & ADRC, Atlanta, Georgia
  - Medical Research Health and Education Foundation, Inc, Columbus, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Josephson, Wallack, Munshower Neurology, PC, Indianapolis, Indiana
  - McLean Hospital, Belmont, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Hattiesburg Clinic, PA, Hattiesburg, Mississippi
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Empire Neurology, PC, Latham, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Dublin, Ohio
  - Lehigh Center for Clinical Research, LLC, Allentown, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Roper St. Francis Healthcare, North Charleston, South Carolina
  - Senior Adult Specialty Research, Austin, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Clinical Neuroscience Research Association, Inc, Bennington, Vermont
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Neurological, PLLC, Spokane, Washington
- Belgium (8):
  - A.Z. Klina, Brasschaat
  - AZ Sint-Jan Brugge, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Centre Neurologique & de Réadaptation Fonctionnelle, Fraiture
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- Canada (13):
  - Health Research., Kamloops, British Columbia
  - Health Research, West Vancouver, British Columbia
  - True North Clinical Research - Halifax Inc., Halifax, Nova Scotia
  - True North Clinical Research Kentville, Inc, Kentville, Nova Scotia
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - St. Joseph's HC- Parkwood Institute, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Recherches Neuro-Hippocampe Inc., Gatineau, Quebec
  - Recherche Sepmus, Inc., Greenfield Park, Quebec
  - DIEX Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Douglas Hospital Research Centre, Verdun, Quebec
- Finland (3):
  - Terveystalo Kamppi, Helsinki
  - Itä-Suomen yliopisto, Aivotutkimusyksikkö, Kuopio
  - CRST, Clinical Research Services Turku, Turku
- France (9):
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Centre de Recherche Clinique du Gérontopôle - Cité de la Santé, Toulouse, Haute Garonne
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hôpital Gui de Chauliac, Montpellier, Herault
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Nantes - Hopital Nord Laënnec, Nantes, Loire Atlantique
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital des Charpennes, Villeurbanne, Rhone
  - Hôpital Fernand Widal, Paris
- Germany (19):
  - Bezirkskrankenhaus Guenzburg, Gunzburg, Baden-Wurttemberg
  - ISPG - Institut fuer Studien zur Psychischen Gesundheit, Mannheim, Baden-Wurttemberg
  - Nervenfachaerztlichen Gemeinschaftspraxis Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinik Hohe Warte Bayreuth, Bayreuth, Bavaria
  - Institut fuer Schlaganfall- und Demenzforschung (ISD), Munich, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Neuropraxis Muenchen Sued, Unterhaching, Bavaria
  - Neuro Centrum Odenwald, Erbach im Odenwald, Hesse
  - Schwerpunktpraxis fuer Neurologie, Psychiatrie und Klinische Studien, Bielefeld, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Zentrum f. Neurologisch- Psychiatrische Studien und Begutachtung, Siegen, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Kopfzentrum Leipzig, Leipzig, Saxony
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - emovis GmbH, Berlin
  - Neurologie im Tempelhofer Hafen, Berlin
- Italy (8):
  - Ospedale degli Infermi, Ponderano, Biella
  - Azienda Ospedaliera Card. G. Panico, Tricase, Lecce
  - ASST di Monza, Monza, Milano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Fondazione Santa Lucia IRCCS, Roma
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
- Japan (23):
  - Research Site, Obu-shi, Aichi-ken
  - Research Site, Toon-shi, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Otake-shi, Hiroshima
  - Research Site, Amagasaki-shi, Hyōgo
  - Research site, Himeji-shi, Hyōgo
  - Research Site, Himeji-shi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Kita-gun, Kagawa-ken
  - Research Site, Kyoto, Kyoto
  - Research Site, Tsu, Mie-ken
  - Research Site, Nishisonogi, Nagasaki
  - Research Site, Yufu-shi, Oita Prefecture
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Okayama, Okayama-ken
  - Research Site, Tsukuba-gun, Okayama-ken
  - Research Site, Kishiwada-shi, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sennan-shi, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Iwata-shi, Shizuoka
  - Research Site, Shizuoka, Shizuoka
- Netherlands (2):
  - Alzheimer Research Center, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
- Poland (14):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - PALLMED Sp. z o.o., Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Novo-Med Zielinski i wspolnicy Sp. j., Katowice
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Centrum Diagnostyczno - Terapeutyczne "MEDICUS" Sp.z o.o., Lubin
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Neurologiczny NZOZ Centrum Leczenia SM, Plewiska
  - NZOZ "NEURO-KARD", "Ilkowski i Partnerzy" Sp. Partn. Lek., Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - NZOZ "SENIOR" Poradnia Psychogeriatryczna, Sopot
  - Osrodek Badan Klinicznych EUROMEDIS, Szczecin
  - Neuro-Care Gabriela Klodowska, Śląskie
  - mMED Maciej Czarnecki, Warsaw
- Spain (9):
  - Hospital General Universitario de Elche, Elche, Alicante
  - ALTHAIA Hospital Sant Joan de Deu, Manresa, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (4):
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Sahlgrenska Universitetssjukhuset, Mölndal Sjukhus, Mölndal
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (6):
  - Universitären Psychiatrischen Kliniken Basel (UPK), Basel
  - Medizinisches Zentrum MZB Biel, Biel/Bienne
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Civico, Lugano
  - Institut fuer Regenerative Medizin (IREM) der Universitaet Zuerich, Zentrum fuer Praevention und Demenztherapie, Schlieren

REFERENCES:
- [Derived] Burton J, Brothers HM, Hutchison RM, Murphy J, Sun T, Dent G, Curiale G, Kowalski K. Lower baseline amyloid beta burden is associated with greater percent of amyloid beta positron emission tomography reduction and better clinical outcomes in the aducanumab Phase 3 trials ENGAGE and EMERGE in early Alzheimer's disease. J Prev Alzheimers Dis. 2025 Aug;12(7):100202. doi: 10.1016/j.tjpad.2025.100202. Epub 2025 May 24. PMID 40413110
- [Derived] Loomis SJ, Miller R, Castrillo-Viguera C, Umans K, Cheng W, O'Gorman J, Hughes R, Budd Haeberlein S, Whelan CD. Genome-Wide Association Studies of ARIA From the Aducanumab Phase 3 ENGAGE and EMERGE Studies. Neurology. 2024 Feb 13;102(3):e207919. doi: 10.1212/WNL.0000000000207919. Epub 2023 Dec 28. PMID 38165296
- [Derived] Muralidharan KK, Kowalski KG, Tong X, Haeberlein SB, Rajagovindan R, Nestorov I. Characterization of exposure-Clinical Dementia Rating-Sum of Boxes relationship in subjects with early Alzheimer's disease from the aducanumab Phase 3 trials. J Pharmacokinet Pharmacodyn. 2023 Feb;50(1):45-62. doi: 10.1007/s10928-022-09839-3. Epub 2023 Jan 4. PMID 36600109
- [Derived] Salloway S, Chalkias S, Barkhof F, Burkett P, Barakos J, Purcell D, Suhy J, Forrestal F, Tian Y, Umans K, Wang G, Singhal P, Budd Haeberlein S, Smirnakis K. Amyloid-Related Imaging Abnormalities in 2 Phase 3 Studies Evaluating Aducanumab in Patients With Early Alzheimer Disease. JAMA Neurol. 2022 Jan 1;79(1):13-21. doi: 10.1001/jamaneurol.2021.4161. PMID 34807243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 181 investigative sites in the United States, Belgium, Canada, Finland, France, Germany, Italy, Japan, Netherlands, Poland, Spain, Sweden, and Switzerland from 15 September 2015 to 13 July 2018.
Pre-assignment Details: A total of 1643 participants with Alzhiemer's disease were enrolled and randomized in the study. Of these, 1638 participants received the study drug in placebo-controlled (PC) period. After completing PC period, 771 participants entered and dosed in long-term extension (LTE) period and no participants completed the study due to early termination of the study.
Groups:
- Placebo (PC Period): Participants received a maximum of 20 infusions of BIIB037-matching placebo intravenously (IV) in PC period, administered approximately once every 4 weeks for up to approximately 1.5 years.
- BIIB037 Low Dose (PC Period): Participants received a maximum of 20 infusions of BIIB037 low dose IV in PC period, administered approximately once every 4 weeks for up to approximately 1.5 years.
- BIIB037 High Dose (PC Period): Participants received a maximum of 20 infusions of BIIB037 high dose IV in PC period, administered approximately once every 4 weeks for up to approximately 1.5 years.
- BIIB037 Late Start: Low Dose (LTE Period): Following PC period, participants randomized to placebo received BIIB037 low dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
- BIIB037 Late Start: High Dose (LTE Period): Following PC period, participants randomized to placebo received BIIB037 high dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
- BIIB037 Early Start: Low Dose (LTE Period): Following PC period, participants randomized to low dose BIIB037 continued to receive the same dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
- BIIB037 Early Start: High Dose (LTE Period): Following PC period, participants randomized to high dose BIIB037 continued to receive the same dose, IV infusion, approximately every 4 weeks for up to 2 years in LTE period.
Period: Placebo-Controlled Period
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | BIIB037 Late Start: Low Dose (LTE Period) | BIIB037 Late Start: High Dose (LTE Period) | BIIB037 Early Start: Low Dose (LTE Period) | BIIB037 Early Start: High Dose (LTE Period)
Started | 548 | 543 | 547 | 0 | 0 | 0 | 0
Completed | 288 | 291 | 295 | 0 | 0 | 0 | 0
Not Completed | 260 | 252 | 252 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 13 | 20 | 0 | 0 | 0 | 0
Not completed — Change of Treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Consent Withdrawn | 15 | 32 | 26 | 0 | 0 | 0 | 0
Not completed — Death | 5 | 0 | 6 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 2 | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Relocation | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Study Visit Burden | 2 | 8 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 4 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 216 | 194 | 183 | 0 | 0 | 0 | 0
Period: Long-Term Extension Period
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | BIIB037 Late Start: Low Dose (LTE Period) | BIIB037 Late Start: High Dose (LTE Period) | BIIB037 Early Start: Low Dose (LTE Period) | BIIB037 Early Start: High Dose (LTE Period)
Started | 0 | 0 | 0 | 131 (11 PC completers did not enter LTE.) | 132 (14 PC completers did not enter LTE.) | 251 (40 PC completers did not enter LTE.) | 257 (38 PC completers did not enter LTE.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 131 | 132 | 251 | 257
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 2 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Loss of Capacity | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Change of Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Consent Withdrawn | 0 | 0 | 0 | 6 | 7 | 13 | 17
Not completed — Investigator Decision | 0 | 0 | 0 | 2 | 1 | 0 | 1
Not completed — Relocation | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Study Visit Burden | 0 | 0 | 0 | 2 | 0 | 0 | 3
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 1 | 3 | 2
Not completed — Reason not Specified | 0 | 0 | 0 | 119 | 117 | 223 | 231

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population was defined as all randomized participants who had received at least one dose of study treatment (Aducanumab or Placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | Total
Number analyzed (Participants) | 548 | 543 | 547 | 1638
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (7.40) | 70.6 (7.45) | 70.6 (7.47) | 70.7 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 290 | 269 | 284 | 843
  Male | 258 | 274 | 263 | 795
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 1
  Race: Asian | 47 | 39 | 42 | 128
  Race: Black or African American | 1 | 6 | 4 | 11
  Race: White | 431 | 432 | 422 | 1285
  Race: Not Reported Due to Confidentiality Regulations | 67 | 65 | 75 | 207
  Race: Other | 1 | 1 | 3 | 5
  Race: Unknown | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethinicity: Hispanic or Latino | 22 | 22 | 23 | 67
  Ethinicity: Not Hispanic or Latino | 470 | 470 | 461 | 1401
  Ethinicity: Not Reported Due to Confidentiality Regulations | 56 | 51 | 62 | 169
  Ethinicity: Unknown | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score at Week 78
Description: CDR-SB integrates assessments from 3 domains of cognition (memory, orientation, judgment/problem-solving) and 3 domains of function (community affairs, home/hobbies, personal care). Following caregiver interview and systematic patient examination, the rater assigns a score describing the participant's current performance level in each of these domains of life functioning. Prespecified severity anchors range from none = 0, questionable = 0.5, mild = 1, moderate = 2 to severe = 3 (the personal care domain omits the 0.5 score). "Sum of boxes" scoring methodology sums the score for each of the 6 domains and provides a value ranging from 0 to 18 that can change in increments of 0.5 or greater. Higher scores indicate greater disease severity. Mixed model for repeated measures (MMRM) analysis was used to analyze change from baseline in CDR-SB. A positive change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: ITT was defined as all randomized participants who had received at least one dose of study treatment (Aducanumab or Placebo). 'Number of Participants Analyzed' signifies number of participants analyzed in this outcome measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 288 | 290 | 299
score on a scale | 1.74 (0.115) | 1.47 (0.116) | 1.35 (0.115)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group (Placebo, BIIB037 Low Dose, BIIB037 High Dose), difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in CDR-SB as dependent variable and with fixed effects of treatment group, categorical visit, treatment-by-visit interaction, baseline CDR-SB, baseline CDR-SB by visit interaction, baseline MMSE, AD symptomatic medication use at baseline, region, and laboratory ApoE status; Test type: Superiority; p = 0.0901, MMRM; Difference = -0.26, 95% CI 2-sided [-0.569 to 0.041]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); Adjusted mean for each treatment group (Placebo, BIIB037 Low Dose, BIIB037 High Dose), difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in CDR-SB as dependent variable and with fixed effects of treatment group, categorical visit, treatment-by-visit interaction, baseline CDR-SB, baseline CDR-SB by visit; Test type: Superiority; p = 0.0120, MMRM; Difference = -0.39, 95% CI 2-sided [-0.694 to -0.086]

2. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Score at Week 78
Description: The MMSE is a widely used performance-based test of global cognitive status. It consists of 11 tasks that assess orientation, word recall, attention and calculation, language abilities, and visuospatial functions. The scores from the 11 tests are combined to obtain the total score, which ranges from 0 to 30, with lower scores over time indicating increasing cognitive impairment. MMRM analysis was used to analyze change from baseline in MMSE. A negative change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 288 | 293 | 299
score on a scale | -3.3 (0.22) | -3.3 (0.22) | -2.7 (0.21)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group (Placebo, BIIB037 Low Dose, BIIB037 High Dose), difference from Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MMSE as dependent variable and with fixed effects of treatment group, categorical visit, treatment-by-visit interaction, baseline MMSE, baseline MMSE by visit interaction, AD symptomatic medication use at baseline, region, and laboratory ApoE status; Test type: Superiority; p = 0.7578, MMRM; Difference = -0.1, 95% CI 2-sided [-0.65 to 0.48]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0493, MMRM; Difference = 0.6, 95% CI 2-sided [0.00 to 1.13]

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (13 Items) (ADAS-Cog 13) at Week 78
Description: ADAS-Cog13 comprises both cognitive tasks and clinical ratings of cognitive performance. The scale items capture word recall, ability to follow commands, the ability to correctly copy or draw an image, naming, the ability to interact with everyday objects, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure for delayed word recall and concentration/distractibility. The total score ranges from 0 to 85. An increase in score over time indicates increasing cognitive impairment. MMRM analysis was used to analyze change from baseline in ADAS-Cog 13. A positive change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 287 | 289 | 293
score on a scale | 5.162 (0.4049) | 4.461 (0.4074) | 3.763 (0.4036)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group(Placebo,BIIB037 Low Dose,BIIB037 High Dose),difference from Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in ADASCog 13 as dependent variable and with fixed effects of treatment group,categorical visit,treatment-by-visit interaction,baseline ADAS-Cog 13,baseline ADAS-Cog 13 by visit interaction,baseline MMSE,AD symptomatic medication use at baseline,region, and laboratory ApoE status; Test type: Superiority; p = 0.1962, MMRM; Difference = -0.701, 95% CI 2-sided [-1.7649 to 0.3627]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0097, MMRM; Difference = -1.400, 95% CI 2-sided [-2.4596 to -0.3396]

4. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment Version) (ADCS-ADL-MCI) Score at Week 78
Description: The ADCS-ADL-MCI consists of 17 instrumental items (e.g., shopping, preparing meals, using household appliances) and 1 basic item (getting dressed). Ratings reflect caregiver observations about the patient's actual functioning over the previous month and provide an assessment of change in the functional state of the participant over time. The total score ranges from 0 to 53, with lower values over time reflecting functional deterioration. MMRM analysis was used to analyze change from baseline in ADAS-ADL-MCI. A negative change from baseline indicates clinical decline.
Time Frame: Baseline, Week 78
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period)
Number analyzed (Participants) | 283 | 286 | 295
score on a scale | -4.3 (0.38) | -3.5 (0.38) | -2.5 (0.38)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB037 Low Dose (PC Period); Adjusted mean for each treatment group (Placebo, BIIB037 Low dose and BIIB037 High Dose), difference from Placebo,95% CI and p-value at each time point were based on an MMRM model, with change from baseline in ADCSADL-MCI as dependent variable and with fixed effects of treatment group, categorical visit, treatment-by-visit interaction, baseline ADCS-ADL-MCI, baseline ADCS-ADL-MCI by visit interaction, baseline MMSE, AD symptomatic medication use at baseline, region, and laboratory ApoE status; Test type: Superiority; p = 0.1515, MMRM; Difference = 0.7, 95% CI 2-sided [-0.27 to 1.73]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB037 High Dose (PC Period); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0006, MMRM; Difference = 1.7, 95% CI 2-sided [0.75 to 2.74]

ADVERSE EVENTS:
Time Frame: From First Dose to End of Study (up to 4 years)
Description: The safety population was defined as all randomised participants who had received at least one dose of study treatment. In PC period, 1 participant randomized to placebo, inadvertently received 1 or more doses of active treatment (Low Dose) during the PC period. For participants affected, a participant was counted only once within each system organ class/preferred term/study period.
Arm/Group | Placebo (PC Period) | BIIB037 Low Dose (PC Period) | BIIB037 High Dose (PC Period) | BIIB037 Late Start: Low Dose (LTE Period) | BIIB037 Late Start: High Dose (LTE Period) | BIIB037 Early Start: Low Dose (LTE Period) | BIIB037 Early Start: High Dose (LTE Period)
All-Cause Mortality (participants affected / at risk) | 5/547 | 0/544 | 6/547 | 0/131 | 0/132 | 3/251 | 0/257
Serious Adverse Events (participants affected / at risk) | 81/547 | 72/544 | 73/547 | 15/131 | 9/132 | 25/251 | 25/257
Other Adverse Events (participants affected / at risk) | 353/547 | 385/544 | 428/547 | 55/131 | 56/132 | 87/251 | 107/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PC Period) (N=547) | BIIB037 Low Dose (PC Period) (N=544) | BIIB037 High Dose (PC Period) (N=547) | BIIB037 Late Start: Low Dose (LTE Period) (N=131) | BIIB037 Late Start: High Dose (LTE Period) (N=132) | BIIB037 Early Start: Low Dose (LTE Period) (N=251) | BIIB037 Early Start: High Dose (LTE Period) (N=257)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femoral hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Medical device site joint pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Cystitis klebsiella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Human anaplasmosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 1 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Animal attack (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 12 | 9 | 4 | 2 | 1 | 1 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0 | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 | 4 | 2 | 0 | 0 | 0 | 0
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 1 | 5 | 8 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dementia alzheimer's type (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Guillain-barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sensorimotor disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Superficial siderosis of central nervous system (Nervous system disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 3 | 2 | 4 | 0 | 1 | 2 | 2
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropsychiatric symptoms (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spermatic cord cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PC Period) (N=547) | BIIB037 Low Dose (PC Period) (N=544) | BIIB037 High Dose (PC Period) (N=547) | BIIB037 Late Start: Low Dose (LTE Period) (N=131) | BIIB037 Late Start: High Dose (LTE Period) (N=132) | BIIB037 Early Start: Low Dose (LTE Period) (N=251) | BIIB037 Early Start: High Dose (LTE Period) (N=257)
Diarrhoea (Gastrointestinal disorders) | 29 | 38 | 42 | 3 | 7 | 9 | 6
Nausea (Gastrointestinal disorders) | 27 | 29 | 31 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 37 | 27 | 34 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 91 | 71 | 89 | 6 | 7 | 18 | 19
Upper respiratory tract infection (Infections and infestations) | 41 | 42 | 38 | 8 | 2 | 13 | 11
Urinary tract infection (Infections and infestations) | 36 | 39 | 29 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 62 | 59 | 73 | 13 | 7 | 15 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 17 | 34 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 38 | 42 | 8 | 3 | 9 | 10
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 37 | 86 | 106 | 18 | 11 | 12 | 21
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 12 | 138 | 183 | 23 | 31 | 11 | 22
Dizziness (Nervous system disorders) | 43 | 42 | 55 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 84 | 109 | 107 | 10 | 13 | 20 | 19
Superficial siderosis of central nervous system (Nervous system disorders) | 14 | 51 | 71 | 13 | 17 | 4 | 10
Anxiety (Psychiatric disorders) | 21 | 30 | 19 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 15 | 16 | 28 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 28 | 29 | 23 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 24 | 33 | 4 | 4 | 7 | 14

LIMITATIONS AND CAVEATS:
The study was halted prematurely based on a prespecified futility analysis and not based on safety concerns. Participants discontinued due to study termination are included in "Reason not Specified" category in participant flow tables above.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information.PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT02484547/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02484547/SAP_001.pdf